CLINICAL TRIAL: NCT02521259
Title: The Correlation Between Anesthetic Depth and the Incidence of Emergence Agitation in Children Undergoing Strabismus Surgery
Brief Title: Anesthetic Depth and the Incidence of Emergence Agitation in Children Undergoing Strabismus Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, LEE YEA JI, clinical professor, Seoul National University Bundang Hospital
Other Study IDs: B-1503-289-004
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Strabismus
Keywords: anesthetic depth; emergence agitation
MeSH Terms: conditions — Strabismus; Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- low Bispectral index (BIS) group: BIS range under 40
  Interventions: Device: BIS
- normal BIS group: BIS range from 40 to 60
  Interventions: Device: BIS

INTERVENTIONS:
Device: BIS — BIS monitoring provides the patient's depth of consciousness, enables us to monitor safe, optimal anesthesia for each patient.

SUMMARY:
This study evaluates the association between the depth of general anesthesia and the occurrence of emergence agitation (EA). The investigators hypothesized that optimal level of anesthetic depth could decrease the incidence of EA in children undergoing strabismus surgery compared to the deep level of anesthetic depth.

DETAILED DESCRIPTION:
EA is characterized by dissociated state of consciousness, in which the children are inconsolable, irritable, uncooperative, thrashing, crying, moaning or incoherent.

Several predisposing factors for EA include post-operative pain, rapid emergence from general anesthesia, use of volatile anesthetics, type and site of operation (usually head & neck surgeries), agitation on induction, airway obstruction, hyperthermia or hypothermia.

The effect of anesthetic depth on the EA has rarely been evaluated in pediatric population, even though postoperative delirium or postoperative cognitive dysfunction (POCD)corresponds to the EA identically.

In this study, the concentration of anesthetics was not managed on purpose to lower the BIS score. Patients were allocated to each group based on the result of average BIS score during the operation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 3 and 5 years
* American Society of Anesthesiologists physical status I or II

Exclusion Criteria:

* American Society of Anesthesiologists physical status over III,
* any disease that could affect mental status
* pre-existing forehead wound

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients, aged between 3 and 5 years, scheduled for strabismus surgery
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: HYO SEOK NA, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, department of Anesthesia and pain, Seongnam, Gyenggo-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Bispectral Index (BIS) Group: Bispectral index (BIS) range from 40 to 60
  BIS: BIS monitoring provides the patient's depth of consciousness, enables us to monitor safe, optimal anesthesia for each patient.
Period: Overall Study
Arm/Group | Normal Bispectral Index (BIS) Group | Low Bispectral Index (BIS) Group
Started | 35 | 33
Completed | 34 | 28
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Bispectral Index (BIS) Group | Normal BIS Group | Total
Number analyzed (Participants) | 28 | 34 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 34 | 62
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 13 | 16 | 29
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: the Pediatric Anesthesia Emergence Delirium (PAED) Score
Description: Evaluating the Pediatric Anesthesia Emergence Delirium (PAED) score 3 times at the post-anesthetic care unit (PACU): when participant arrived at PACU, measure the PAED score (from 0 to 20; the higher score indicates the severer emergenct agitation) immediately and if the score is 10 or over 10, give the participant Fentanyl 1mcg/kg. Repeat checking the PAED score 2 times more with 15 minutes interval.
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low Bispectral Index (BIS) Group | Normal BIS Group
Number analyzed (Participants) | 28 | 34
score on a scale
  T1 (on arrival PACU) | 12.5 (5.0) | 11.4 (5.4)
  T2 (15 minutes after T1) | 6.5 (1.3) | 5.4 (3.4)
  T3 (15 minutes after T2) | 3.2 (2.0) | 3.4 (2.5)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every 6 months.
Description: In this study, the concentration of inhalational agent was conventional in both group. We didn't manage the concentation intentionally to make BIS lower than 40 even in Low BIS Group. There were no adverse event and/or serious adverse event.
Arm/Group | Low Bispectral Index (BIS) Group | Normal BIS Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/34
Other Adverse Events (participants affected / at risk) | 0/28 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No